CLINICAL TRIAL: NCT03999177
Title: Pilot Usability and Feasibility Testing on Kinect-Enhanced Training System for Lymphatic Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19-00222; 1R01CA214085 (NIH)
Record Dates: First submitted 2019-06-24; First posted 2019-06-26 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Breast Cancer; Lymphedema
MeSH Terms: conditions — Breast Neoplasms; Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Kinect-TOLF prototype (Experimental)
  Interventions: Behavioral: Kinect-TOLF Training System

INTERVENTIONS:
Behavioral: Kinect-TOLF Training System — This system will teach patients to perform the lymphatic exercises correctly. Like playing the video games, patients follow the avatar model in the video to perform the lymphatic exercises. The Kinect system can automatically detect whether a user is performing the set of lymphatic exercises correctly in real time and provide instantaneous feedback to the user, thus enhancing patients' self-efficacy to perform the lymphatic exercises correctly. Patients will be asked to conduct two types of usability testing: heuristic evaluation and end-user testing.

SUMMARY:
Correct performance of therapeutic lymphatic exercises has the potential to relieve lymphedema symptoms and optimize limb volume and lymph fluid level, in turn to improve breast cancer survivors' quality of life and reduce the risk of lymphedema. Kinect-TOLF (Kinect-Enhanced The-Optimal-Lymph-Flow Training System) is an innovative intelligent Kinect-enhanced training system to teach patients to perform the lymphatic exercises correctly. The Kinect-TOLF training system is not a medical device but a computer/mobile and motion-sensor program that helps patients to perform the lymphatic exercises correctly. The Kinect system can automatically detect whether a user is performing the set of lymphatic exercises correctly in real time and provide instantaneous feedback to the user, thus enhancing patients' self-efficacy to perform the lymphatic exercises correctly. The goal of the proposed project is to evaluate the usability and feasibility of Kinect-TOLF.

ELIGIBILITY:
Inclusion Criteria:

* Women who have received surgical treatment for breast cancer (Stage I-III), including mastectomy, lumpectomy, sentinel lymph node biopsy (SLNB), SLNB plus lymph node dissection or axillary lymph nodes dissection
* Report any persistent or intermittent pain or lymphedema symptoms in the ipsilateral upper limb or body at least 8 weeks after surgery, that is, beyond the expected period of healing
* May or may not have had neoadjuvant therapy or adjuvant therapy of chemotherapy or radiation
* Have history or no history of lymphedema or have or not been treated for lymphedema;
* Able to speak and understand English since the proposed usability testing is designed to only test the English version of the intervention.
* Women willing to come to the NYU Perlmutter Cancer Center for the research visit.

Exclusion Criteria:

* Women diagnosed with breast cancer but did not undergo surgical treatment as breast surgery and removal of lymph nodes are the major treatment-related risk factors for lymphedema;
* Known metastatic disease (Stage IV), recurrence of cancer, or lymphedema due to cancer recurrence, or other bulk disease in the thoracic or cervical regions;
* Women with renal or heart failure, cardiac pacemaker or defibrillator, artificial limbs, or pregnant women as accurate measurement of body mass index (BMI) may not be possible with an impedance device according to the manufactures.

Ages: 21 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
The Perceived Ease of Use and Usefulness | 12 Months
  a tool to evaluate users' acceptance of a new information system with a strong reliability for perceived usefulness and perceived ease of use [49-50]. We used the modified eight-items with 5-point Likert Scales ranging from 2 (strongly agree) to -2 (strongly disagree) for this usability evaluation.
The Post Study System Usability Questionnaire | 12 Months
  originally is a 19-item survey instrument developed at IBM to assess user satisfaction with system usability on a scale ranging from 1 (strongly agree) to 7 (strongly disagree). We will use the modified 13-item tool from the original survey that focus on system usefulness and information quality (Lewis 1995). The survey consists of three subscales accounted for 87 percent of the total variance: system usefulness, information quality and interface quality. The overall reliability of the survey was 0.97, and ranged from 0.91 to 0.96 for the three subscales.

CONTACTS AND LOCATIONS:
Overall Officials: Mei Fu, PhD, RN, FAAN, Principal Investigator — New York Langone Medical Center
Locations (1):
- NYU Langone Health, New York, New York, United States

REFERENCES:
- [Derived] Fu MR, McTernan ML, Qiu JM, Ko E, Yazicioglu S, Axelrod D, Guth A, Fan Z, Sang A, Miaskowski C, Wang Y. The Effects of Kinect-Enhanced Lymphatic Exercise Intervention on Lymphatic Pain, Swelling, and Lymph Fluid Level. Integr Cancer Ther. 2021 Jan-Dec;20:15347354211026757. doi: 10.1177/15347354211026757. PMID 34160294